CLINICAL TRIAL: NCT03483714
Title: Muscle Activation Characteristics During Spinal Manipulation in Healthy and Low Back Pain Participants
Status: Completed | Type: Observational
Sponsor: University of Denver (Other)
Responsible Party: Principal Investigator, Stuart Currie, Principle Investigator, University of Denver
Other Study IDs: LSM
Record Dates: First submitted 2018-03-11; First posted 2018-03-30 (Actual); Last update posted 2018-03-30 (Actual); Status verified 2018-03

CONDITIONS: Back Pain
Keywords: Manipulation; Spinal; electromyography; kinetics; kinematic
MeSH Terms: conditions — Back Pain | interventions — Manipulation, Spinal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy Participants: Spinal manipulation
  Interventions: Procedure: Spinal Manipulation
- Acute Low back pain participants: Spinal Manipulation
  Interventions: Procedure: Spinal Manipulation
- Chronic low back pain participants: Spinal Manipulation
  Interventions: Procedure: Spinal Manipulation

INTERVENTIONS:
Procedure: Spinal Manipulation — HVLA (High Velocity Low Amplitude) spinal manipulation directed at the lumbar spine and sacroiliac (SI) joints

SUMMARY:
To characterize muscle activity through electromyography (EMG) of the lumbar spine during high velocity, low amplitude (HVLA) spinal manipulation according to parameters of practitioner contact (location, applied force) in healthy participants and two categories of low back pain participants.

ELIGIBILITY:
Inclusion Criteria:

* male and female participants ages 18 to 55 years old

Exclusion Criteria:

Active Worker's Compensation claim related to low back pain episode Active personal injury case related to low back pain episode Currently taking muscle relaxers, steroids, or narcotics

* Body mass index > 30 kg/m2
* Active cancer process
* Active infection
* Pregnancy
* High risk of osteoporosis assessed using the World Health Organization Fracture Risk Assessment Tool (included in submission)
* Osteogenic conditions (see screening questionnaire)
* Premature menopause
* Latex Allergies
* Lumbar spine or pelvic surgery
* Past spinal trauma producing spinal fracture

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: community sample
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2011-02-01 (Actual); Primary Completion 2015-11-05 (Actual); Study Completion 2015-11-05 (Actual)

PRIMARY OUTCOMES:
Muscle Response | During spinal manipulation at the time of testing
  Muscle activity of the lumbar spinal musculature as measured by both surface and indwelling electromyography. Total response expressed as a percentage of muscles "on".
Muscle Activity Onset Delay | During spinal manipulation at the time of testing
  Muscle activity of the lumbar spinal musculature as measured by both surface and indwelling electromyography. Time delay between the manipulation force and the muscle activity

CONTACTS AND LOCATIONS:
Overall Officials: Bradley S Davidson, PhD, Principal Investigator — University of Denver
Locations (1):
- University of Denver, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Currie SJ, Myers CA, Krishnamurthy A, Enebo BA, Davidson BS. Methods of Muscle Activation Onset Timing Recorded During Spinal Manipulation. J Manipulative Physiol Ther. 2016 May;39(4):279-87. doi: 10.1016/j.jmpt.2016.03.001. Epub 2016 Apr 9. PMID 27072513
- [Result] Currie SJ, Myers CA, Durso C, Enebo BA, Davidson BS. The Neuromuscular Response to Spinal Manipulation in the Presence of Pain. J Manipulative Physiol Ther. 2016 May;39(4):288-93. doi: 10.1016/j.jmpt.2016.02.011. Epub 2016 Apr 6. PMID 27059250
- [Result] Myers CA, Enebo BA, Davidson BS. Optimized prediction of contact force application during side-lying lumbar manipulation. J Manipulative Physiol Ther. 2012 Nov-Dec;35(9):669-77. doi: 10.1016/j.jmpt.2012.10.010. PMID 23206961